CLINICAL TRIAL: NCT00957333
Title: Effects of Ketamine on Human Bladders and Its Possible Mechanisms
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DOH98-NNB-1049
Record Dates: First submitted 2009-08-03; First posted 2009-08-12 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2010-11

CONDITIONS: Cystitis
Keywords: ketamine; bladder dysfunction; bladder mucosa; mechanisms
MeSH Terms: conditions — Cystitis | interventions — Ketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1.Urine 2.Blood 3.Biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- case: ketamine + Cystitis
  Interventions: Other: ketamine

INTERVENTIONS:
Other: ketamine

SUMMARY:
This study is aimed to evaluate the relationship between ketamine abused and bladder dysfunction and its possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* Cystitis (the clinicians ruled out the causes of bacterial infection)
* Frequent micturition
* The clinicians are willing to sign the ICF

Exclusion Criteria:

* Suffers from the urinary system disease, is not suitable to carry on the urinary bladder biopsy sampling
* Suffers from other diseases, doctor recognized that is not suitable to carry on the sampling
* The clinicians are not willing to sign the ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruei-Ming Chen, PhD, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Case: ketamine + Cystitis
  ketamine
Period: Overall Study
Arm/Group | Case
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Case
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 27
Region of Enrollment [Number; unit: participants]
  Taiwan | 44

OUTCOME MEASURES:

1. Primary Outcome: Substance Abuse Situation Record
Description: Substance abuse situation record: ketamine
Time Frame: 1 day
Measure: Mean (Full Range); unit: years
Arm/Group | Case
Number analyzed (Participants) | 44
years | 2 [0.5 to 5]

2. Secondary Outcome: Urinary Bladder Capacity
Time Frame: 1 day
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Case
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No